CLINICAL TRIAL: NCT01081301
Title: Living With Hope: Developing a Psychosocial Supportive Program for Rural Older Women Caregivers of Spouses With Advanced Cancer
Brief Title: Living With Hope Program for Rural Women Caregivers
Acronym: LWH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Wendy Duggleby, Professor, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BEH 08-186; 184186 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Advanced Cancer
Keywords: hope; quality of life; caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Living with Hope Program (Experimental): Receive Living with Hope Program
  Interventions: Behavioral: Living with Hope Program

INTERVENTIONS:
Behavioral: Living with Hope Program — The LWHP consists of the LWH film featuring caregivers of patients with advanced cancer describing their hope and a hope activity "Stories of the Present". Following viewing of the video with trained research assistants (RAs), (without discussion) the RA's will instruct the subjects to take 5 minutes at the end of the day and write about their thoughts, challenges and what gave them hope over a 2 week time period. Subjects can choose to use a journal, a computer or audiotape their journals.

SUMMARY:
Family caregivers of terminally ill persons describe hope as inner strength that will help them continue caregiving. Our research team has developed and pilot tested a Living with Hope Program (LWHP) for caregivers of family members with advanced cancer, with the goal of fostering hope and improving quality of life (www.usask.ca/nursing /research/livingwithhope). The caregivers involved in our pilot test found the LWHP easy to use and we found some evidence to suggest that the program may have increased their hope and improved their quality of life. We would like to further develop and test the LWHP by finding out more about how and how long it might work. We believe it will improve the quality of life of active and bereaved older rural women of persons with advanced cancer and may decrease the number of prescriptions and doctor visits over one year. Since rural women caring for persons with advanced cancer seem to have the least hope, we want to focus on them first before including other caregivers in our research. Two hundred rural women caring for a person with advanced cancer will be asked to take part in this study. Their feelings of control, loss and grief, quality of life and hope will be measured over a year. The numbers of time they visit their physician and how many prescriptions they have over the year will also be collected. This study will contribute to the refinement of a Living with Hope Program that may improve quality of life and personal health of older rural women caring for their spouse with advanced cancer and those who subsequently become bereaved.

DETAILED DESCRIPTION:
1. Background: The research team has developed and pilot tested a Living with Hope Program (LWHP) for caregivers of family members with advanced cancer. The LWHP includes viewing an award winning Living with Hope video followed by writing a daily journal for two weeks. The pilot test findings suggested that the LWHP is an acceptable and feasible intervention for use by family caregivers. Although the LWHP shows promise in potentially increasing hope and quality of life, further testing and development is needed. Questions remain as to: a) what are the mechanisms through which the LWHP affects outcomes and b) how long it is effective?
2. Purpose: The overall purpose of this time series mixed method study is the further development and testing of the LWHP by:

   1. Determining the mechanisms of the LWHP by testing the LWHP conceptual model in which self-efficacy and loss and grief are hypothesized intervening variables for changes in hope, and subsequently quality of life among rural women caring for persons with advanced cancer. In the LWHP model we hypothesize that administration of the LWHP will improve self-efficacy and decrease feelings of loss and grief. This will lead to a positive influence on the proximal outcome of hope and the distal outcome of quality of life.
   2. Exploring the longitudinal effects of the LWHP on hope, quality of life and health services utilization among older rural women caring for spouses with advanced cancer. We want to determine if the LWHP has benefits beyond what was found in the pilot. The team will compare baseline scores of hope and quality of life to scores after the LWHP over time and health services utilization (one year prospective number of physician visits and prescriptions compared to the year before the LWHP). This study is unique, as it will follow caregivers over a one-year period. As approximately 50% of these caregivers will become bereaved one month after study enrolment; rather than dropping these caregivers from the study, the team felt that retaining these subjects would add to the understanding of hope, quality of life and health care utilization among caregivers by continuing to follow them through bereavement. Thus, patterns of hope, quality of life and health care services utilization will be delineated over time for active and bereaved caregivers.
3. Research Plan: Using a time-series embedded mixed method design, baseline measures were collected from 122 rural women caring for a person who has advanced cancer. Data collection began January 2009 in 4 sites: Saskatoon Cancer Agency, Alan Blair Cancer Agency, Sunrise Health Region and Regina/Qu'Appelle Health Region. Data collection in Alberta started July 2010 through Alberta Health Services Community Cancer Clinics, and in September 2010 through a mail out through the Alberta Cancer Registry. In January 2011 subjects were enrolled through a mail out through the Saskatchewan Cancer Registry. Subjects who consented to participate in the full study received the LWHP. Subjects were then post tested on the variables at 1 and 2 weeks, 3, 6 and 12 months. Journal entries were copied and transcribed.
4. Data Analysis: Path Analysis will be used to test the model post LWHP at 1 and 2 weeks. Two-factor ANCOVA will determine patterns over time and Cortazzi's narrative analysis will be used to analyze the subjects journals completed as part of the LWHP.
5. Significance: This study will contribute to the refinement of the Living with Hope Program that may improve quality of life and personal health of older rural women caring for their spouse with advanced cancer and those who subsequently become bereaved. The findings will also increase our understanding of the factors influencing hope, quality of life and health in a vulnerable, understudied population that is increasing in numbers with the aging of Canada's population. Family care giving is what sustains patients at the end of life, and with changing demographics and diminishing resources there is a potential that every Canadian will be an informal caregiver at some time. Effective psychosocial supportive interventions, such as the LWHP are critical for their support and well-being.

ELIGIBILITY:
Inclusion Criteria:

* caring for a person who is diagnosed with advanced cancer, c) home address is outside of metropolitan areas.

Exclusion Criteria:

* caring for a person with advanced cancer and dementia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy D Duggleby, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Duggleby W, Holtslander L, Kylma J, Duncan V, Hammond C, Williams A. Metasynthesis of the hope experience of family caregivers of persons with chronic illness. Qual Health Res. 2010 Feb;20(2):148-58. doi: 10.1177/1049732309358329. PMID 20065303
- [Background] Duggleby WD, Williams AM. Living with hope: developing a psychosocial supportive program for rural women caregivers of persons with advanced cancer. BMC Palliat Care. 2010 Mar 26;9:3. doi: 10.1186/1472-684X-9-3. PMID 20346156
- [Derived] Duggleby W, Williams A, Holstlander L, Cooper D, Ghosh S, Hallstrom LK, McLean RT, Hampton M. Evaluation of the living with hope program for rural women caregivers of persons with advanced cancer. BMC Palliat Care. 2013 Oct 9;12(1):36. doi: 10.1186/1472-684X-12-36. PMID 24106841

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Saskatchewan, the Palliative Care Admission team in Regina Qu'Appelle Health Region and nurses at the Saskatchewan Cancer Agency also identified potential participants. In Alberta, the Alberta Health Services Cancer Care and Community Cancer Clinics in rural communities also identified potential participants.
Pre-assignment Details: Exclusion criteria were a) women who were cognitively impaired as determined by the recruitment team at the site, b) women otherwise unable to participate, in the opinion of the recruitment team and c) women caring for a family member who has a diagnosis of advanced cancer as well as dementia.
Groups:
- Living With Hope Program: Receive Living with Hope Program
  Living with Hope Program : The LWHP consists of the LWH film featuring caregivers of patients with advanced cancer describing their hope and a hope activity "Stories of the Present". Following viewing of the video with trained research assistants (RAs), (without discussion) the RA's will instruct the subjects to take 5 minutes at the end of the day and write about their thoughts, challenges and what gave them hope over a 2 week time period. Subjects can choose to use a journal, a computer or audiotape their journals.
Period: Overall Study
Arm/Group | Living With Hope Program
Started | 36
Completed | 22
Not Completed | 14
Not completed — Bereaved | 3
Not completed — Too busy | 5
Not completed — Patient too ill | 2
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Living With Hope Program
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 36
Herth Hope Index [Mean (Standard Deviation); unit: units on a scale] — The Herth Hope Index provides a summative hope score and scores for three sub-scales of hope: a) temporality and future, b) positive readiness and expectancy, and c) interconnectedness. It is a 12 item likert response scale (1-4) with summative scores ranging from 12-48, with a higher score denoting greater hope. It has reported reliability (test-retest r=0. 91, p<0. 05) and validity (concurrent validity, r=0. 84, p<.0 05; criterion, r=. 92, p< 0.05; divergent, r=-.73, p<0. 05).
  units on a scale | 37.79 (5.97)
General Self-Efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — This likert type scale has 10 items which produces a total perceived general self-efficacy score. Responses are made on a 4 point scale. Scores range from 10 to a maximum score of 40; the higher scores the higher participant feelings of self-efficacy. The GSES has been found to be a reliable and valid measure in many populations and countries and has been used in a study of hope and family caregivers of women with breast cancer. Reliability ranges from r=0.76 to r=0.90 and criterion related reliability was r=0.80, p<0.05.
  units on a scale | 31.1 (3.94)
Short Form Health Survey Version 2 - Mental Health [Mean (Standard Deviation); unit: units on a scale] — The SF-12v2 was developed as a shorter yet valid alternative to the SF 36 as a measure of quality of life. The SF-12v2 produces a physical health component summary score (PCS), and a mental health component summary score (MCS), but not a total summary score. Scores range from 0 (poor health) to 100 (perfect health). The SF-12v2 physical summary and mental health summary scores correlate very highly (r=0.95 and 0.96 respectively) with the SF-36 and have reported test-retest reliability of r=0.89 and 0.76 respectively.
  units on a scale | 43.59 (5.35)
Short Form Health Survey Version 2 - Physical Health [Mean (Standard Deviation); unit: units on a scale] — The SF-12v2 was developed as a shorter yet valid alternative to the SF 36 as a measure of quality of life. The SF-12v2 produces a physical health component summary score (PCS), and a mental health component summary score (MCS), but not a total summary score. Scores range from 0 (poor health) to 100 (perfect health). The SF-12v2 physical summary and mental health summary scores correlate very highly (r=0.95 and 0.96 respectively) with the SF-36 and have reported test-retest reliability of r=0.89 and 0.76 respectively.
  units on a scale | 45.17 (3.87)
Non-Death Revised Grief Experience Inventory [Mean (Standard Deviation); unit: units on a scale] — The NDRGEI is a 22-item scale measuring four domains of the grief experience for people who are not bereaved (item examples are in brackets): 1) existential concerns (e.g. "I feel lost and helpless"), 2) depression (e.g. "I cry easily"), 3) guilt (e.g. "I have feelings of guilt"), and 4) distress (e.g. "My arms and legs feel very heavy"). Responses are scored on a 6-point scale, ranging from slight disagreement to strong agreement, with a higher total score indicating more grief and loss. The Non-Death Revised Grief Experience Inventory has a minimum score of 22 and a maximum score of 132.
  units on a scale | 72.82 (23.92)

OUTCOME MEASURES:

1. Primary Outcome: Herth Hope Index
Description: The Herth Hope Index is a 12 item (1-4 point) Likert scale that delineates three sub-scales of hope: a) temporality and future, b) positive readiness and expectancy, and c) interconnectedness. These three subscales are consistent with descriptions of hope by caregivers in the preliminary work completed by the research team. The subscales also include measures of relationships and spirituality that are considered factors that influence hope. Summative scores range from 12-48, with a higher score denoting greater hope.
Time Frame: Baseline, 1week, 2 weeks, 3, 6 and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living With Hope Program [Baseline] | Living With Hope Program [Day 7] | Living With Hope Program [Day 14] | Living With Hope Program [3 Months] | Living With Hope Program [6 Months] | Living With Hope Program [12 Months]
Number analyzed (Participants) | 36 | 35 | 33 | 31 | 26 | 22
units on a scale | 37.79 (5.97) | 39.74 (4.96) | 39.06 (6.05) | 38.17 (5.22) | 39.34 (4.96) | 40.53 (5.2)
Statistical Analysis 1: Comparison: Living With Hope Program [Baseline] vs Living With Hope Program [12 Months]; Generalized estimating equations were used to determine change in patterns of the Herth Hope Index over time (Day 7, 14 and 3, 6, and 12 months) compared to baseline. The advantage of utilizing general estimating equations was that it effectively increases the sample size (increasing power) and estimated more robust standard errors by taking into account the repeated measures and adjusting for covariates; Test type: Superiority or Other; p < 0.05, ANOVA — The p-value were not adjusted for multiple comparisons and a p-value of 0.05 was used for statistical significance; Modified version of ANOVA as it overcomes the shortcoming of the ANOVA model by taking into account unbalanced data and repeated measures

2. Secondary Outcome: SF12 Mental Health
Description: The SF12 was developed to be a shorter yet valid alternative to the SF 36 as a measure of quality of life. The SF12 measures 7 concepts: Physical functioning, role limitations due to physical health problems, bodily pain, general healthy vitality, social functioning, role limitations due to emotional problems and mental health. It produces a physical component summary score (PCS), and a mental health component summary score (MCS). Scores range from 0 (poor health) to 100 (perfect health).
Time Frame: baseline, 1 and 2 wks, 3, 6 and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Living With Hope Program [Baseline]: Baseline Measure
- Living With Hope Program [Day 7]: Day 7 Receive Living with Hope Program
  Living with Hope Program : The LWHP consists of the LWH film featuring caregivers of patients with advanced cancer describing their hope and a hope activity "Stories of the Present". Following viewing of the video with trained research assistants (RAs), (without discussion) the RA's will instruct the subjects to take 5 minutes at the end of the day and write about their thoughts, challenges and what gave them hope over a 2 week time period. Subjects can choose to use a journal, a computer or audiotape their journals.
- Living With Hope Program [Day 14]: Day 14 Receive Living with Hope Program
  Living with Hope Program : The LWHP consists of the LWH film featuring caregivers of patients with advanced cancer describing their hope and a hope activity "Stories of the Present". Following viewing of the video with trained research assistants (RAs), (without discussion) the RA's will instruct the subjects to take 5 minutes at the end of the day and write about their thoughts, challenges and what gave them hope over a 2 week time period. Subjects can choose to use a journal, a computer or audiotape their journals.
- Living With Hope Program [3 Months]: 3 months Receive Living with Hope Program
  Living with Hope Program : The LWHP consists of the LWH film featuring caregivers of patients with advanced cancer describing their hope and a hope activity "Stories of the Present". Following viewing of the video with trained research assistants (RAs), (without discussion) the RA's will instruct the subjects to take 5 minutes at the end of the day and write about their thoughts, challenges and what gave them hope over a 2 week time period. Subjects can choose to use a journal, a computer or audiotape their journals.
- Living With Hope Program [6 Months]: 6 months Receive Living with Hope Program
  Living with Hope Program : The LWHP consists of the LWH film featuring caregivers of patients with advanced cancer describing their hope and a hope activity "Stories of the Present". Following viewing of the video with trained research assistants (RAs), (without discussion) the RA's will instruct the subjects to take 5 minutes at the end of the day and write about their thoughts, challenges and what gave them hope over a 2 week time period. Subjects can choose to use a journal, a computer or audiotape their journals.
- Living With Hope Program [12 Months]: 12 months Receive Living with Hope Program
  Living with Hope Program : The LWHP consists of the LWH film featuring caregivers of patients with advanced cancer describing their hope and a hope activity "Stories of the Present". Following viewing of the video with trained research assistants (RAs), (without discussion) the RA's will instruct the subjects to take 5 minutes at the end of the day and write about their thoughts, challenges and what gave them hope over a 2 week time period. Subjects can choose to use a journal, a computer or audiotape their journals.
Arm/Group | Living With Hope Program [Baseline] | Living With Hope Program [Day 7] | Living With Hope Program [Day 14] | Living With Hope Program [3 Months] | Living With Hope Program [6 Months] | Living With Hope Program [12 Months]
Number analyzed (Participants) | 36 | 35 | 33 | 31 | 26 | 22
units on a scale | 43.59 (5.35) | 45.27 (5.66) | 44.15 (6.40) | 45.57 (5.76) | 44.52 (5.66) | 47.15 (5.36)
Statistical Analysis 1: Comparison: Living With Hope Program [Baseline] vs Living With Hope Program [12 Months]; Generalized estimating equations were used to determine change in patterns of SF-12v2 Mental health scores over time (Day 7, 14 and 3, 6, and 12 months) compared to baseline. The advantage of utilizing general estimating equations was that it effectively increases the sample size (increasing power) and estimated more robust standard errors by taking into account the repeated measures and adjusting for covariates; Test type: Superiority or Other; p < 0.05, ANOVA — The p-value were not adjusted for multiple comparisons and a p-value of 0.05 was used for statistical significance; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: General Self-Efficacy Score (GSES)
Description: The scale consists of 10 items with responses from 1-4. The higher the Scores on the General Self Efficacy Scale (which has a range from 10 - 40), indicate higher participant feelings of self-efficacy. The General Self Efficacy Scale was chosen as a measure for this study because it has been found to be a reliable and valid measure in many populations.
Time Frame: Baseline, 1week, 2 weeks, 3, 6 and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Living With Hope Program [Baseline]: Receive Living with Hope Program
  Living with Hope Program : The LWHP consists of the LWH film featuring caregivers of patients with advanced cancer describing their hope and a hope activity "Stories of the Present". Following viewing of the video with trained research assistants (RAs), (without discussion) the RA's will instruct the subjects to take 5 minutes at the end of the day and write about their thoughts, challenges and what gave them hope over a 2 week time period. Subjects can choose to use a journal, a computer or audiotape their journals.
Arm/Group | Living With Hope Program [Baseline] | Living With Hope Program [Day 7] | Living With Hope Program [Day 14] | Living With Hope Program [3 Months] | Living With Hope Program [6 Months] | Living With Hope Program [12 Months]
Number analyzed (Participants) | 36 | 35 | 33 | 31 | 26 | 22
units on a scale | 31.1 (3.94) | 33.04 (4.03) | 32.44 (4.41) | 32.63 (3.64) | 33.2 (3.74) | 33.2 (4.44)
Statistical Analysis 1: Comparison: Living With Hope Program [Baseline] vs Living With Hope Program [12 Months]; Generalized estimating equations were used to determine change in patterns of General Self Efficacy Scale scores over time (Day 7, 14 and 3, 6, and 12 months) compared to baseline. The advantage of utilizing general estimating equations was that it effectively increases the sample size (increasing power) and estimated more robust standard errors by taking into account the repeated measures and adjusting for covariates; Test type: Superiority or Other; p < 0.05, ANOVA — The p-value were not adjusted for multiple comparisons and a p-value of 0.05 was used for statistical significance; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Non-Death Revised Grief Experience Inventory
Description: The Non-Death Revised Grief Experience Inventory measures grief that is not associated with the death of a person. It is a 22-item scale measuring four domains (existential concerns, depression, tension and guilt, and physical distress) of the grief experience. Responses are scored on a 6-point scale, ranging from slight disagreement to strong agreement, with higher total score indicating more grief and loss. The Non-Death Revised Grief Experience Inventory has a minimum score of 22 and a maximum score of 132.
Time Frame: Baseline, 1week, 2 weeks, 3, 6 and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living With Hope Program [Baseline] | Living With Hope Program [Day 7] | Living With Hope Program [Day 14] | Living With Hope Program [3 Months] | Living With Hope Program [6 Months] | Living With Hope Program [12 Months]
Number analyzed (Participants) | 36 | 35 | 33 | 31 | 26 | 22
units on a scale | 72.82 (23.92) | 71.75 (24.13) | 70.22 (22.23) | 73.26 (23.6) | 64.63 (25.59) | 66.29 (24.43)
Statistical Analysis 1: Comparison: Living With Hope Program [Baseline] vs Living With Hope Program [12 Months]; Generalized estimating equations were used to determine change in patterns of Non Death Revised Grief Experience Inventory scores over time (Day 7, 14 and 3, 6, and 12 months) compared to baseline. The advantage of utilizing general estimating equations was that it effectively increases the sample size (increasing power) and estimated more robust standard errors by taking into account the repeated measures and adjusting for covariates; Test type: Superiority or Other; p > 0.05, ANOVA — The p-value were not adjusted for multiple comparisons and a p-value of 0.05 was used for statistical significance; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: SF12: Physical Health
Description: as for outcome 2
Time Frame: Baseline, 1week, 2 weeks, 3, 6 and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living With Hope Program [Baseline] | Living With Hope Program [Day 7] | Living With Hope Program [Day 14] | Living With Hope Program [3 Months] | Living With Hope Program [6 Months] | Living With Hope Program [12 Months]
Number analyzed (Participants) | 36 | 35 | 33 | 31 | 26 | 22
units on a scale | 45.17 (3.87) | 44.36 (4.47) | 45.56 (5.05) | 45.1 (5.31) | 43.98 (4.67) | 43.37 (5.28)
Statistical Analysis 1: Comparison: Living With Hope Program [Baseline] vs Living With Hope Program [12 Months]; Generalized estimating equations were used to determine change in patterns of SF-12v2 Physical health scores over time (Day 7, 14 and 3, 6, and 12 months) compared to baseline. The advantage of utilizing general estimating equations was that it effectively increases the sample size (increasing power) and estimated more robust standard errors by taking into account the repeated measures and adjusting for covariates; Test type: Superiority or Other; p < 0.05, ANOVA — The p-value were not adjusted for multiple comparisons and a p-value of 0.05 was used for statistical significance; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Living With Hope Program [Baseline] | Living With Hope Program [Day 7] | Living With Hope Program [Day 14] | Living With Hope Program [3 Months] | Living With Hope Program [6 Months] | Living With Hope Program [12 Months]
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/35 | 0/33 | 0/31 | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 0/36 | 0/35 | 0/33 | 0/31 | 0/26 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes